CLINICAL TRIAL: NCT05336916
Title: (Cost)Effectiveness of Blended and UnguideD DeliverY of Mindfulness-based Cognitive Therapy Versus Care as Usual for Cancer Patients: BUDDY Project
Brief Title: Effectiveness of Blended and Unguided Delivery of Mindfulness-based Cognitive Therapy for Cancer Patients
Acronym: BUDDY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL73117.091.20
Record Dates: First submitted 2022-03-23; First posted 2022-04-20 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: Cancer; Mindfulness-based Cognitive Therapy (MBCT); Blended intervention; eHealth
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blended MBCT (Experimental): The blended MBCT consists of four 2,5 hour group sessions through videoconference (session 1, 3, 5 and 8), taught by experienced mindfulness trainers. The other sessions (2, 4, 6 and 7) are delivered online and are individual. Mindfulness trainers will provide online feedback to participants for these sessions. The sessions include meditation exercises, psycho-education, and group discussion. In addition to the sessions, participants are instructed to do daily home practice 45 minutes a day. The regular MBCT program was adapted to fit the needs of the target group and, for instance includes psycho-education about grief and cancer-related fatigue.
  Online sessions were built around a specific theme. Participants are provided with information, audio files of meditations, and recording assignments around the theme of the session through a personal, secure webpage. The sessions look appealing and persuasive technologies such as reminders and videos are used.
  Interventions: Behavioral: Buddy
- Unguided online MBCT (Experimental): Participants in the unguided online arm receive access to the 8 online mindfulness sessions (same intervention as blended MBCT arm), but no mindfulness trainer will be involved.
  Each online session was built around a specific theme, for instance automatic pilot, communication or self-care. Participants are provided with information, audio files of meditations, and recording assignments around the theme of the session through a personal, secure webpage. Participants are encouraged to read the information and do the assigned meditations and recording assignments within one week. The sessions will look appealing and persuasive technologies such as reminders and video's will be used.
  Interventions: Behavioral: Buddy
- Treatment As Usual (No Intervention): Not offered the mindfulness program, treatment as usual

INTERVENTIONS:
Behavioral: Buddy — Mindfulness-based Cognitive Behavioural Therapy
  Arms: Blended MBCT; Unguided online MBCT

SUMMARY:
Rationale: Approximately one in three cancer patients and survivors experience significant psychological distress. Previous research has shown that mindfulness-based interventions such as mindfulness-based cognitive therapy (MBCT) can help reduce distress among cancer patients. However, MBCT typically takes place in face-to-face group sessions, which are not easily accessible to many cancer patients. Blended therapist-assisted (combination of group sessions and individual online sessions) and unguided online MBCT interventions may address this problem, however, research on effectiveness of these interventions is missing.

Objective: This three-armed, randomized controlled trial (RCT) evaluates the effectiveness and cost-effectiveness of blended therapist-assisted (blended MBCT) and unguided individual internet-based MBCT (online MBCT) compared to treatment-as-usual (TAU) for cancer patients. Secondly, consolidation of treatment effects is studied up to nine months post-treatment. Thirdly, possible working mechanisms and effect moderators are studied.

Study design: The current study is a RCT with three arms (blended MBCT, online MBCT and TAU) with assessments at baseline (T0), mid-treatment, post-treatment (T1) and 3 months follow-up (T2). At 3 months follow-up (T2), patients in the TAU arm will be crossed over to blended MBCT or online MBCT (random allocation). Uncontrolled follow-up assessments will be conducted at 6 (T3) and 9 months (T4) follow-up.

Study population: 254 adults (>18 years) who have or have had a cancer diagnosis (any stage/any type) will be randomized.

Intervention: Patients will be randomly assigned with a 1:1:1 ratio to one of three groups: (1) blended MBCT: patients will be invited to a blended therapist-assisted MBCT program, consisting of 8 weekly sessions (4 online group meetings, 4 online sessions with therapist assistance, and an online silent day), in addition to TAU; (2) online MBCT: patients will be invited to an individual internet-based MBCT program without assistance from a therapist, that consists of 8 weekly sessions and a silent day, in addition to TAU; (3) TAU: patients receive usual care, which can be medical, psychological or paramedical care, except mindfulness interventions.

Main study parameters/endpoints: Primary outcome is the difference in Hospital Anxiety and Depression Scale (HADS) total scores between patients in the blended MCBT and TAU arms and between the online MCBT and TAU arms post-treatment (T1).

DETAILED DESCRIPTION:
About one in three cancer patients experience significant levels of psychological distress, requiring intervention from a health professional. Unfortunately, however, many cancer patients experiencing psychological symptoms do not receive treatment.

Effective psychological treatments for cancer patients are available. Evidence for the effectiveness of mindfulness-based interventions (MBIs) such as Mindfulness-based Stress Reduction (MBSR) and Mindfulness-Based Cognitive Therapy (MBCT) in oncology has rapidly increased. MBIs have beneficial effects on depression symptoms, anxiety, fear of cancer recurrence and fatigue. Also, preliminary results indicate that MBIs are cost-effective in cancer care.

However, there are known patient-reported barriers to engaging in face-to-face psychological interventions, such as investment of time, stigma, reluctance to return to the hospital, and indirect costs. In contrast, internet-based interventions are easily accessible and save travelling time. Evidence of over 100 trials suggests that internet-based treatments can be as effective as face-to-face treatments for psychiatric and somatic conditions. MBIs are also being delivered via Internet, but research on internet-based MBIs (eMBIs) has been mostly conducted in the general population.

Studies on the effectiveness of eMBIs in cancer patients are scarce. Our team conducted the first RCT comparing group MBCT and individual internet-based MBCT with TAU in patients with cancer. Therapist-assisted individual internet-based MBCT was similar to group MBCT in terms of treatment protocol, but took place individually and was guided one-on-one by a therapist on a weekly basis. Results indicated that both group MBCT and individual internet-based MBCT were significantly effective in reducing psychological distress in cancer patients compared to TAU. Moreover, both interventions significantly increased secondary quality-of-life outcomes with small to moderate effect sizes. Patients further improved over the course of the 9 months post-treatment, with patients who were less conscientious and less mindful at baseline benefitting more from therapist-assisted individual internet-based MBCT than group MBCT. Cost-effectiveness analyses demonstrated dominance of both interventions compared to TAU, indicating both higher quality of life and lower societal costs. In short, individual internet-based MBCT rendered MBCT much more accessible for cancer patients without compromising intervention efficacy or societal costs.

However, the proportion of patients receiving a lower dosage of MBCT than intended was substantially higher in individual internet-based MBCT than in group MBCT and although cost-effective, the individual internet-based MBCT proved to be resource intensive in terms of therapist assistance. Moreover, patients mentioned lack of peer support and the asynchronous communication with their therapist as important disadvantages of individual internet-based MBCT. Consequently, there is room to improve individual internet-based MBCT prior to implementation to ensure adherence and scalability.

To improve adherence and scalability, the investigators have developed two new versions of the effective online MBCT program with therapist assistance in a co-creation process together with relevant stakeholders. To improve adherence, a blended therapist-assisted MBCT (blended MBCT) was developed, combining four online group sessions with a therapist with four individual therapist-assisted online sessions. Furthermore, to improve scalability, unguided individual internet-based MBCT (online MBCT), which is similar to the previously studied individual internet-based MBCT protocol but without therapist guidance was also developed. As adherence to unguided interventions often is lower than intended, persuasive technology known to improve adherence was included, such as reminders and virtual coaches.

The current study primarily aims to investigate the effectiveness and cost-effectiveness of blended MBCT and online MBCT in comparison to treatment-as-usual (TAU) in a randomized controlled trial (RCT). Secondly, the aim is to test the consolidation of treatment effects up to nine months post-treatment. Thirdly, the investigators want to investigate working mechanisms and treatment effect moderators, to address how these programs work, and for whom.

The aim is to include 254 patients who were diagnosed with cancer (any stage, any tumor). After baseline assessment, patients will be randomized to the blended MBCT, unguided online MBCT or TAU (1:1:1 ratio). Outcome assessment for the RCT will occur at baseline (T0), immediately post-treatment (T1; primary endpoint) and three months follow-up (T2). Patients participating will also receive follow-up questionnaires at 6 months (T3) and 9 months (T4) post-treatment. At week 5 of both interventions (and at the same time during TAU), patients will be invited to complete a mid-treatment assessment, to look at working mechanisms. At 3 months follow-up (T2), patients in TAU will be randomized to the blended MBCT or unguided online MBCT.

ELIGIBILITY:
Inclusion Criteria:

1. A cancer diagnosis, any tumor or stage
2. Computer literacy and internet access
3. Good command of the Dutch language
4. Willingness to participate in either MBCT intervention

Exclusion Criteria:

1. Previous participation in MBSR or MBCT (>4 sessions)
2. Severe psychiatric comorbidity that warrants acute treatment (psychosis, mania, severe personality disorders, suicidal thoughts)
3. Alcohol or drug dependence
4. Severe cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Difference in Hospital Anxiety and Depression Scale (HADS) total scores between patients in the Blended MBCT arm and TAU, and between patients in the Online MBCT arm and TAU | 1 week post-treatment
  The HADS is a 14-item questionnaire measuring distress. Items are scored on a 0-3 scale that are summed to obtain a distress total score (range 0-42). Higher scores represent more distress.

SECONDARY OUTCOMES:
Difference in Hospital Anxiety and Depression Scale (HADS) total scores between patients in the Blended MBCT arm and TAU, and between patients in the Online MBCT arm and TAU | 3, 6 and 9 months post-treatment
  The HADS is a 14-item questionnaire measuring distress. Items are scored on a 0-3 scale that are summed to obtain a distress total score (range 0-42). Higher scores represent more distress.
Difference in Fear of Cancer Recurrence Inventory (FCRI) severity subscale scores between patients in the Blended MBCT arm and TAU, and between patients in the Online MBCT arm and TAU | 1 week post-treatment and 3, 6 and 12 months post-treatment
  The 9-item Fear of Cancer Recurrence Inventory severity subscale assesses fear of cancer recurrence on a 5-point Likert scale ranging from 0 (not at all or never) to 4 (a great deal or all the time). Higher scores indicate higher levels of FCR.
Difference in Checklist Individual Strength (CIS)- Fatigue scores between patients in the Blended MBCT arm and TAU, and between Online MBCT arm and TAU | 1 week post-treatment and 3, 6 and 12 months post-treatment
  The 8-item CIS-Fatigue Severity measures the patient's fatigue levels over the past 2 weeks on a 7-point scale, with higher scores indicating higher levels of fatigue.
Difference in Rumination and Reflection Questionnaire (RRQ) rumination subscales scores between patients in the Blended MBCT arm and TAU, and between Online MBCT arm and TAU | 1 week post-treatment and 3, 6 and 12 months post-treatment
  Rumination will be measured using the rumination 12-item subscale of the Rumination and Reflection Questionnaire. Items are scored on a five-point rating scale, with higher scores indicating more rumination.
Difference in Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) scores between patients in the Blended MBCT arm and TAU, and between patients in the Online MBCT arm and TAU | 1 week post-treatment and 3, 6 and 12 months post-treatment
  The 24-item Five Facet Mindfulness Questionnaire Short Form assesses mindfulness skills and consists of five subscales: observing, describing, acting with awareness, non-judging of inner experience and non-reactivity to inner experience. Items are scored on a five-point rating scale (1 = rarely true, 5 = always true). Higher scores are indicative of someone who is more mindful in their everyday life.
Difference in Decentering subscale of the Experiences Questionnaire scores between patients in the Blended MBCT arm and TAU, and between patients in the Online MBCT arm and TAU | 1 week post-treatment and 3, 6 and 12 months post-treatment
  The 11-item Decentering subscale of the Experiences Questionnaire measures the ability to observe one's thoughts and feelings as temporary, objective events in the mind. Participants rate items on a 5-point Likert scale (1 = never to 5 = always). Higher scores indicate greater decentering ability.
Difference in Self-Compassion Scale Short Form (SCS-SF) scores between patients in the Blended MBCT arm and TAU, and between patients in the Online MBCT arm and TAU | 1 week post-treatment and 3, 6 and 12 months post-treatment
  The Self-compassion Scale-Short Form is a 12-item self-report measure that is used to measure people's capacity for self-compassion. Items are scored on a five-point Likert scale (0 = 'Almost never' to 5 = 'Almost always') to record how often you behave kindly and caringly towards yourself in difficult life situations. Higher scores reflect higher levels of self-compassion.
Difference in Mental Health Continuum-Short Form (MHCSF) scores between patients in the Blended MBCT arm and TAU, and between patients in the Online MBCT arm and TAU | 1 week post-treatment and 3, 6 and 12 months post-treatment
  The 14-item MHCSF measures positive mental health, consisting of three subscales: 1) emotional well-being, 2) psychological well-being, and 3) social well-being. Items assess the frequency with which respondents experience each symptom of positive mental health on a 6-point Likert scale ranging from 0 "never" to 5 "everyday" Higher scores indicate greater levels of positive well-being.
Difference in EuroQol-5D-5L (EQ-5D) index scores between patients in the Blended MBCT arm and TAU, and between patients in the Online MBCT arm and TAU | 1 week post-treatment and 3, 6 and 12 months post-treatment
  The EQ-5D is a generic instrument comprising five domains with five levels: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D index is obtained by applying predetermined weights to the five domains. This index gives a societal-based global utility score of the participant's health status on a scale with 0 (death) and 1 (perfect health)
Difference in the Trimbos/iMTA questionnaire for Costs associated with Psychiatric illness (TiC-P) between patients in the Blended MBCT arm and TAU, and between patients in the Online MBCT arm and TAU | 1 week post-treatment and 3, 6 and 12 months post-treatment
  The Trimbos/iMTA questionnaire for Costs associated with Psychiatric illness (TiC-P) will be used to collect information on direct healthcare use (e.g. general practitioner, mental healthcare and hospital day care visits) and paid and informal work-related productivity losses. Higher scores indicate greater healthcare use and productivity losses.
Engagement with the intervention will be measured with Twente Engagement with Ehealth Technologies Scale (TWEETS) among participants in the blended and online MCBT arms | 1 week post-treatment
  The TWEETS consists of 9 items, divided over 3 subscales: behavioural engagement, cognitive engagement and affective engagement. On a scale of 1 to 5, participants indicate the extent to which they agree with statements such as "I think I will be able to use this [technology] as often as needed [to achieve my goals]" (behavioural engagement), "this [technology] will motivate me to [goal of the technology]" (cognitive engagement) or " I think I will enjoy using this [technology]" (affective engagement).

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after the collection of the primary outcome
Access Criteria: Approval of proposed purpose for data access

REFERENCES:
- [Derived] Badaghi N, Kwakkenbos L, Prins J, Donders R, Kelders S, Speckens A. Randomized Controlled Trial of Group-Blended and Individual-Unguided Online Mindfulness-Based Cognitive Therapy to Reduce Psychological Distress in People With Cancer. Psychooncology. 2025 Sep;34(9):e70286. doi: 10.1002/pon.70286. PMID 40968786
- [Derived] Badaghi N, van Kruijsbergen M, Speckens A, Vile J, Prins J, Kelders S, Kwakkenbos L. Group, Blended and Individual, Unguided Online Delivery of Mindfulness-Based Cognitive Therapy for People With Cancer: Feasibility Uncontrolled Trial. JMIR Form Res. 2024 Feb 21;8:e52338. doi: 10.2196/52338. PMID 38381493
- [Derived] Badaghi N, van Kruijsbergen M, Prins J, Kelders S, Cillessen L, Compen F, Donders R, Kwakkenbos L, Speckens A. Effect of blended and unguided online delivery of mindfulness-based cognitive therapy versus care as usual on distress among cancer patients and survivors: protocol for the three-arm parallel randomized controlled buddy trial. BMC Psychol. 2023 Jan 25;11(1):21. doi: 10.1186/s40359-023-01052-2. PMID 36698197